CLINICAL TRIAL: NCT03509454
Title: PeRsOnalising Treatment Of Diabetic Nephropathy: From Albuminuria to Multidimensional Characterisation of Diabetic Nephropathy - a Cross-sectional Study
Brief Title: PeRsOnalising Treatment Of Diabetic Nephropathy:
Acronym: PROTON
Status: Completed | Type: Observational
Sponsor: Peter Rossing (Other)
Responsible Party: Sponsor-Investigator, Peter Rossing, Professor, MD, DMsc, Steno Diabetes Center Copenhagen
Organization: Steno Diabetes Center Copenhagen (Other)
Other Study IDs: 36000
Record Dates: First submitted 2018-04-10; First posted 2018-04-26 (Actual); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Complications; Diabetic Nephropathies
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Complications; Diabetic Nephropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood urine and fecal samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Type 1 DM, Normo albuminuric: Type 1 diabetics with no history of albumnuria (UACR < 30 mg/g in 2 out of 3 consecutive samples)
- Type 1 DM, Micro albuminuric: Type 1 diabetics with history of micro albumnuria (UACR 30-299 mg/g in 2 out of 3 consecutive samples)
- Type 1 DM, Macro albuminuric: Type 1 diabetics with history of macro albumnuria (UACR 30-299 mg/g in 2 out of 3 consecutive samples)
- Healthy subjects: Subjects with no history of diabetes, other diseases or intake of medicine which in the judgement of the investigator could affect the results, specifically renal, cardiovascular or inflammatory/infectious diseases should be considered for exclusion.

SUMMARY:
Background: Today diabetic nephropathy is a frequent, and the most lethal and costly complication of diabetes. Although treating blood pressure with agents blocking renin angiotensin system has improved outcome, the prognosis is still poor and no new interventions have been successful during the past decade. There is an urgent need for discovery of new pathways behind the development and progression of diabetic nephropathy as well as of biomarkers which can identify subjects at risk of developing adverse events. Objective: By using a multidimensional 'omics' approach, we aim to search for novel proteins, metabolites and pathways that will point to the putative new mechanisms which underlie the early renal decline.

Design: Cross-sectional study, with long-term register-based follow-up. Study population: 160 patients with type 1 diabetes recruited from Steno Diabetes Center Copenhagen stratified based on stage of diabetic kidney disease, and 50 healthy non-diabetic controls. Endpoints: Primary endpoint: Glycocalyx thickness, assessed as perfused boundary region. Secondary endpoints: Gut microbiome characterisation and markers of gastrointestinal inflammation, autonomic and periphery neuropathy, urine and plasma Flow Cytometry Analysis (FACS), metabolomics and proteomics in plasma and urine, and other potential biomarkers.

DETAILED DESCRIPTION:
Design: Cross-sectional study, with long-term register-based follow-up. Study population: 160 patients with type 1 diabetes recruited from Steno Diabetes Center Copenhagen stratified based on stage of diabetic kidney disease, and 50 healthy non-diabetic controls. Endpoints: Primary endpoint: Glycocalyx thickness, assessed as perfused boundary region. Secondary endpoints: Gut microbiome characterisation and markers of gastrointestinal inflammation, autonomic and periphery neuropathy, urine and plasma Flow Cytometry Analysis (FACS), metabolomics and proteomics in plasma and urine, and other potential biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 diabetes
* Written informed consent must be provided before participation
* Male or female patients >18 years of age with a diagnosis of type 1 diabetes (WHO criteria)
* Persistent urinary albumin creatinine ratio (UACR) assessed from EPJ (Electronic Patient Journal):
* < 30 mg/g in 2 out of 3 consecutive samples (normoalbuminuria)
* 30 - 299 mg/g in 2 out of 3 consecutive samples (microalbuminuria)
* ≥ 300 mg/g in 2 out of 3 consecutive samples (macroalbuminuria) - at least 30 with concurrent eGFR < 60 ml/min/1.73m2

  2. Control subjects without diabetes
* Written informed consent must be provided before participation.
* Male or female patients >18 years of age without a diagnosis of diabetes (assessed by Hb1Ac, haemoglobin and creatinine)

Exclusion Criteria: (Both subjects with and without diabetes)

* Non-diabetic kidney disease as indicated by medical history and/or laboratory findings
* Renal failure (eGFR<15 ml/min/1.73m2), dialysis or kidney transplantation
* Change in RAAS blocking treatment during the last month
* Treatment with antibiotics during the last 2 month
* Pregnancy or breastfeeding (urine HCG is performed on all fertile women)
* Patients who, in the judgement of the investigator, is incapable to participate
* For controls: Other diseases or intake of medicine which in the judgement of the investigator could affect the results, specifically renal, cardiovascular or inflammatory/infectious diseases should be considered for exclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 160 patients with type 1 diabetes and different stages of diabetic nephropathy (50 with normoalbuminuria; 50 with microalbuminuria; and 60 with macroalbuminuria -including at least 30 with concurrent estimated Glomerular Filtration Rate (eGFR) < 60 ml/min/1.73m2) compared to 50 healthy non-diabetic controls.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
The microvascular function by estimating the glycocalyx thickness | 2019
  Glycocalyx thickness assessed as perfused boundary region by a hand-hold camera (GlycoCheck)

SECONDARY OUTCOMES:
Gut microbiome | 2019
  Characterisation of the gut microbiota and markers of gastrointestinal inflammation
Urine and plasma Flow Cytometry Analysis (FACS) | 2019
  cell types related to inflammation
Metabolomics in plasma | 2019
  metabolite risk score in plasma
Metabolomics in urine | 2019
  metabolite risk score in urine
proteomics in urine | 2019
  proteomic risk score in urine
proteomics in plasma | 2019
  proteomic risk score in plasma
Autonomic neuropathy | 2019
  beat to beat variation (R-R test) upon Deep breathing
peripheral neuropathy | 2019
  vibration perception threshold

CONTACTS AND LOCATIONS:
Overall Officials: peter Rossing, Study Chair — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center, Gentofte Municipality, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No